CLINICAL TRIAL: NCT01817023
Title: Multicenter Phase III Study of Intensity-modulated Radiotherapy Alone Compared to Intensity-modulated Radiotherapy Combined Chemotherapy for Lower Risk Locally Advanced Nasopharyngeal Carcinoma
Brief Title: The Role of Concurrent Chemotherapy for Lower Risk Locally Advanced Nasopharyngeal Carcinoma(NPC) in the Era of IMRT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jun-Lin Yi, MD, Vice chairman， Department of Radiation Oncology, Cancer hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CH-HN-003
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2020-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; current chemotherapy; intensity-modulated radiotherapy; low-risk
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin

STUDY DESIGN:
Who Masked: Investigator
Masking Description: central investigator organization digital randomize
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RT alone (Experimental): SIB-IMRT was given to the patients with a regimen of 69.96Gy-73.92Gy to the gross target volume, 60Gy to the high risk clinical target volume, 50Gy to the low risk clinical target volume
  Interventions: Radiation: SIB-IMRT
- CCRT group (Active Comparator): SIB-IMRT was given to the patients with regimen of 69.96Gy-73.92Gy to the gross target volume, 60Gy to the high risk clinical target volume, 50Gy to the low risk clinical target volume and cisplatin 100mg/m2 was given at d1, d22,d43 during radiotherapy.
  Interventions: Radiation: SIB-IMRT; Drug: Cisplatin

INTERVENTIONS:
Radiation: SIB-IMRT — SIB-IMRT was given to the patients with regimen of 69.96Gy-73.92Gy to the gross target volume, 60Gy to the high risk clinical target volume, 50Gy to the low risk clinical target volume
Drug: Cisplatin — Cisplatin 100mg/m2 was delivered at d1,d22 and d43 to the CCRT group patients during radiotherapy.
  Arms: CCRT group

SUMMARY:
The purpose of this study is to verify that simultaneous integrated boost IMRT (SIB-IMRT) alone is non-inferior to SIB-IMRT combined with concurrent chemotherapy for low-risk locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
* There were several randomized clinical trials confirmed that concurrent chemoradiotherapy (CCRT) is superior to radiotherapy (RT)alone for locally advanced NPC, most of the patients in the trials were treated with conventional radiotherapy technique.
* As the new technique of IMRT used more and more in the clinical practice, the role of concurrent chemoradiotherapy (CCRT) seems blurred, in two of Hongkong phaseIII studies(NPC9901/9902), half of the patients were treated by 3-dimensional conformal radiotherapy (3DCRT)/IMRT,the results showed that there were no significant different in terms of overall survival between RT alone and CCRT groups. Furthermore, several large sample size retrospective studies from China, showed that there were no advantage of CCRT over RT alone when treated by SIB-IMRT.
* In an analysis of who will benefit from CCRT,( Lin, et.al, IJROBP,2004; 60:156-164), the author divided the locally advanced NPC patients into two groups, with the high-risk group defined as patients met at least one of following criteria: nodal size >6 cm, (2) supraclavicular node metastasesN3, T4N2 and multiple neck node metastases with 1 node >4cm.
* Based on these information, we hypothesize that, for low-risk locally advanced NPC patients, there may no need CCRT under SIB-IMRT treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological proven non-keratin nasopharyngeal carcinoma
* AJCC 7th edition stage III/IVM0, without any one of following factors: node size >6cm;supraclavicular metastasis node; T4N2; multiple neck node metastases with 1 node >4 cm
* Life expectancy≥6 months
* Adequate renal function, defined as follows: Serum creatinine < 2 x institutional upper limit of normal(ULN) within 2 weeks prior to registration or creatinine clearance rate (CCr) ≥ 50 ml/min within 2 weeks prior to registration determined by 24- hour collection or estimated by Cockcroft-Gault formula: CCr male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dl) x (72)] CCr female = 0.85 x (CCrmale)
* The following assessments are required within 2 weeks prior to the start of registration: Na, K, Cl, glucose, Ca, Mg, and albumin

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years; noninvasive cancers (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible) are permitted even if diagnosed and treated < 3 years ago
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Severe, active co-morbidity
* Treatment planning does not meet the requirement of prescription dose.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2013-04; Primary Completion 2019-07-30 (Actual); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years
  according to the recruitment, a interrim analysis will done in July, 2019, if there is inferior finding of RT alone group, the study will premature terminate

SECONDARY OUTCOMES:
Acute and late toxicities | 5years
  * compare the acute radiation and chemotherapy-related toxicities during treatment course
  * compare late toxicities after treatment
3 year Progression-free survival (PFS) | 5year
  to compare the 3years PFS between the IMRT alone and IMRT with concurrent chemoradiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Li Gao, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (6):
- China (6):
  - Department of nasopharyngeal carcinoma, Cancer hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Department of Radiation oncology, Cancer hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Tongji hospital, Huazhong University of Science & Technology, Wuhan, Hubei
  - Jiangxi province cancer hospital, Nanchang, Jiangxi
  - Cancer hospital, Chinese Academy of Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: No